CLINICAL TRIAL: NCT03067168
Title: A Multicenter, Double Blinded, Randomized Controlled Trial of Levator Muscle Blocks Following Posterior Colporrhaphy Surgery to Reduce Post-operative Pain.
Brief Title: A Trial of Levator Muscle Blocks Following Posterior Colporrhaphy Surgery to Reduce Post-operative Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christ Hospital (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Carson T. Kaeser, MD, Fellow in Female Pelvic Medicine and Reconstructive Surgery, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCH# 15-02
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will not know if they received an injection of bupivacaine or placebo, i.e., normal saline after completion of surgery. The surgeon, as well as any investigator or study personnel, will be blinded to injection type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine Arm (Active Comparator): The subjects of this arm will receive an injection of 5mL of 0.5% bupivacaine, 1-2 cm deep to the surface of the vaginal epithelium into the levator ani muscle, puborectalis. A second injection of 5mL of 0.5% bupivacaine, 1-2 cm deep to the surface of the vaginal epithelium will be repeated on the same side, approximately 2-3 cm cephalad of the first injection at the iliococcygeus muscle. These 2 injections will then be repeated on the contralateral side.
  Interventions: Drug: Bupivacaine
- Placebo Arm (Placebo Comparator): The subjects of this arm will receive an injection of 5mL of 0.9% normal saline, 1-2 cm deep to the surface of the vaginal epithelium into the levator ani muscle, puborectalis. A second injection of 0.9% normal saline, 1-2 cm deep to the surface of the vaginal epithelium will be repeated on the same side, approximately 2-3 cm cephalic from first injection at the iliococcygeus muscle. These 2 injections will then be repeated on the contralateral side.
  Interventions: Drug: normal saline 0.9%

INTERVENTIONS:
Drug: Bupivacaine — 5 mL of 0.5% bupivacaine will be injected into 2 locations bilaterally.
  Other Names: Marcaine
  Arms: Bupivacaine Arm
Drug: normal saline 0.9% — 5 mL of 0.9% normal saline will be injected into 2 locations bilaterally.
  Other Names: Saline
  Arms: Placebo Arm

SUMMARY:
To determine if levator muscle block with bupivacaine improves postoperative pain control relative to placebo controls among women undergoing prolapse surgery involving a posterior colporrhaphy. Improvement is defined as no less than a 25% lower total pain score on a ten point numerical pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Any woman over the age of 18 years with a capacity to give informed consent who are undergoing vaginal prolapse surgery including a posterior colporrhaphy may be included in the study.

Exclusion Criteria:

* Any woman who is a non-English speaker, does not have ability to provide consent, has a cardiac arrhythmia, liver disease, myasthenia gravis, bleeding diathesis or adverse reaction / allergy to anesthetic will be excluded. Women that are also having vaginal mesh excisions at the time of prolapse repair or those that will undergo subsequent surgery in the follow up period will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients that are eligible would be undergoing vaginal prolapse surgery including posterior colporrhaphy, therefore would need to have a vagina to be enrolled in this study
Enrollment: 128 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement in pain, scored on a 10 point numerical pain scale. | 1 year
  Improvement is defined as a 25% or lower total pain score on a ten point numerical pain scale compared to placebo.

SECONDARY OUTCOMES:
Postoperative care satisfaction scores, graded with a post-operative survey. | 1 year
  Improvement in satisfaction is defined as an overall satisfaction score of 20% or more on the post-operative survey compared to placebo.
Measure of morphine equivalents used in patients postoperatively. | 1 year
  A reduction in opiate use is defined as a 20% reduction in total number of morphine equivalents used between study cohorts.
Length of hospital stay measured in hours. | 1 year
  Length, in hours, of hospital stay between study cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Carson T Kaeser, MD, Principal Investigator — The Christ Hospital
Locations (3):
- United States (3):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The Christ Hospital, Cincinnati, Ohio
  - The University of Toledo, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaeser CT, Rothenberger R, Zoorob D, Whiteside JL. Bupivacaine Use After Posterior Colporrhaphy to Reduce Postoperative Pain: A Multicenter, Double-Blinded, Placebo-Controlled, Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2022 Feb 1;28(2):72-76. doi: 10.1097/SPV.0000000000001082. PMID 34171880